CLINICAL TRIAL: NCT06612281
Title: Evaluation of Gixam's Performance in a FIT Negative Population
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jubaan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL-1015
Record Dates: First submitted 2024-09-09; First posted 2024-09-25 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Adenoma; Colorectal Cancer (CRC); Colorectal Cancer (CRC) Screening
Keywords: Microbiome; Spectral signature; Artificial intelligence
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: All subjects enrolled will undergo the same study procedures and assessments in the following order: FIT, Gixam, and colonoscopy. Gixam is an investigational medical device determined by the FDA to be a nonsignificant risk device. Colonoscopy is the ground-truth (Gixam outcome is compared to colonoscopy findings). Gixam performance will be evaluated and reported per FIT outcome (the primary efficacy endpoint is sensitivity and specificity in a FIT negative population).
Masking Description: Participant and physician performing colonoscopy will be masked to FIT and Gixam test outcome until colonoscopy procedure us completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm (Experimental): All participants will undergo the same study procedures: FIT, Gixam, and colonoscopy
  Interventions: Device: colorectal cancer (CRC) screening; Diagnostic Test: colorectal cancer screening; Procedure: Colonoscopy after bowel cleansing

INTERVENTIONS:
Device: colorectal cancer (CRC) screening — Gixam test
Diagnostic Test: colorectal cancer screening — Fecal Immunochemistry Test (FIT)
Procedure: Colonoscopy after bowel cleansing — Standard of care optical colonoscopy for colorectal cancer screening

SUMMARY:
In the United States, colorectal cancer ranks second to lung cancer as a cause of cancer death and is the third most commonly occurring cancer in both men and women. Colorectal cancer in most cases develops slowly over a period of years, starting with the growth of precancerous polyps on the colon or rectum wall. The slow development of colorectal cancer makes it possible to detect and prevent it entirely by the removal of the precancerous polyps with colonoscopy. To date, there is no screening test, other than colonoscopy, able to detect the precancerous polyps. Gixam is a camera that takes multiple pictures of your tongue and uses artificial intelligence software to predict the presence of precancerous polyps within your colon or rectum that may eventually become cancerous.

The device creates the prediction by comparing the images taken of your tongue with many other images of tongues from healthy patients and patients with a history of precancerous polyps. Patients who have been predicted by Gixam to have precancerous polyps may be more likely to complete colonoscopy at the interval recommended by their physician, potentially reducing the likelihood of developing colorectal cancer.

The purpose of this research study is to test the accuracy of the Gixam device in persons that have received a negative outcome on a Fecal Immunochemical Test (FIT). This study will compare this prediction to the actual findings of your scheduled standard care colonoscopy and allow researchers to evaluate and improve the Gixam system.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 45-85 years.
2. Able to provide a signed informed consent.
3. Scheduled for a screening colonoscopy at the investigation site.

Exclusion Criteria:

1. Undergoing diagnostic colonoscopy for investigation of symptoms.
2. Has undergone colonoscopy within preceding nine (9) years except for a failed colonoscopy due to poor bowel preparation. Failed colonoscopy must have been within the past year and without therapeutic intervention.
3. History of colorectal cancer.
4. Family history of colorectal cancer, defined as having one or more first-degree relatives (parent, sibling, or child) with CRC at any age.
5. Subject has a diagnosis or medical / family history of any of the following conditions, including:

   * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome),
   * Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome"),
   * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis, or Familial Hyperplastic Polyposis.
6. Subject has a diagnosis or personal history of inflammatory bowel disease (IBD) including chronic ulcerative colitis and/or Crohn's disease.
7. Subjects with a disability to extend their tongue.
8. Subjects with tongue piercing.
9. Dental visit in the past 7 days prior to Gixam test.
10. Intake of pro-biotics over the past 3 months pre-Gixam test.
11. Subject has any condition that in the opinion of the Investigator should preclude participation in the study.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety - number of device related adverse events and serious adverse events | Through study completion, up to 30 days
  Number of device related adverse events and serious adverse events
Efficacy - Gixam's sensitivity and specificity | Through study completion, up to 30 days
  Gixam's sensitivity and specificity to predict the presence of colorectal adenoma or sessile serrated lesions (advances and non-advanced) / CRC in a FIT negative population.

CONTACTS AND LOCATIONS:
Locations (1):
- The Oregon Clinic Gastroenterology-East, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://jubaan.com/